CLINICAL TRIAL: NCT06223841
Title: A Clinical Trial of Phase Ib/II to Evaluate Effect of IAP0971 in Patients With Advanced Malignant Tumors
Brief Title: A Clinical Trial to Evaluate Effect of IAP0971 in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IAP0971-202
Record Dates: First submitted 2024-01-05; First posted 2024-01-25 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ib - Dose escalation (Experimental)
  Interventions: Drug: IAP0971
- Phase II - Clinical Exploratory Stage (Experimental)
  Interventions: Drug: IAP0971

INTERVENTIONS:
Drug: IAP0971 — IAP0971 should be subcutaneous injected，q3w

SUMMARY:
This is a Phase Ib/II Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Effectiveness of IAP0971 in Patients with Advanced Malignant Tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 to 75years, male or female.
* 2. Phase Ib:With advanced or metastatic malignant solid tumor confirmed by histopathology, the standard treatment fails, or there is no standard treatment plan, or standard treatment is not applicable at this stage, or the patient refuses the standard treatment, or the investigator evaluates the patient who can benefit from this treatment.
* 3.Phae II: Confirmed by histopathology that it is not feasible to perform complete resection and cannot be connected. Locally advanced (stage IIIB or IIIC) or metastatic (IV) after radical concurrent radiotherapy and chemotherapy Stage) non-small cell lung cancer (NSCLC). Note: For unacceptable radical synchronization/sequencing.Subjects with locally advanced stage IIIB/IIIC of radiotherapy and chemotherapy need to be evaluated by relevant professional doctors. And provide written records to confirm.
* 4.Phae II: Never received systemic anti-tumor therapy for locally advanced or metastatic NSCLC before. Tumor treatment(received adjuvant/neoadjuvant chemotherapy or radical treatment for locally advanced diseases) .Patients with synchronous or sequential radiotherapy and chemotherapy and disease progression occurred after the last treatment ≥6 months).
* 5.Phase II: PD-L1 was positive (TPS≥50%) by IHC, and the patient was immunohistochemical. Epidermal growth factor receptor (EGFR) and anaplasticlymphomakinase (ALK) were negative.
* 6. At least one measurable tumor lesion per RECIST 1.1 (solid tumors).
* 7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. 7. The estimated survival time is ≥3 months.8.Adequate organ function: Hematological system (No blood transfusion or hematopoietic stimulating factor therapy within 14 days) Absolute neutrophil count (ANC) ≥ 1.5 × 109/L White blood cell count (WBC) ≥ 3.0 × 109/L Platelets (PLT) ≥ 75 × 109/L Hemoglobin (Hb) ≥ 90 g/L Hepatic function Total bilirubin (TBIL) ≤ 3 × ULN Alanine aminotransferase (ALT) ≤ 3 × ULN; Aspartate aminotransferase (AST) ≤ 3 × ULN; Renal function Creatinine clearance (Ccr) (only calculated if creatinine > 3 × ULN) ≥ 50 mL/min (calculated according to Cockcroft-Gault formula, see Appendix 7 for formula) Coagulation function Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN International normalized ratio (INR) ≤ 1.5 × ULN.
* 8. Expected survival time of more than 3 months.
* 9. Eligible patients of childbearing potential (men and women) must agree to use a reliable method of contraception (hormonal or barrier method or abstinence, etc.) with their partners during the trial and for at least 90 days after study drug administration; female patients of childbearing potential (see Appendix 8 for definition) must have a negative blood or urine pregnancy test 7 days before the first administration.
* 10. Eligible patients with fertility (male and female) must agree that during and at the end of the trial.Use reliable contraceptive methods (hormones or screens) with their partners for at least 6 months after taking the drug.Obstacle law or abstinence); Blood of female patients of childbearing age within 7 days before the first use of the study drug.The pregnancy test must be negative.
* 11.Subjects must be informed of the study prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

* 1.Phase II: Pathohistologically confirmed with small cell lung cancer components, or sarcomatoid lesions.
* 2. Phase II : Previous immunotherapy, including immune checkpoint inhibitors (such as PD-1/PD-L1 antibody, anti-CTLA-4 antibody, etc.), immune checkpoint agonist (such as:ICOS, CD40, CD137, GITR, OX40 antibody, etc.), immune cell therapy, etc.
* 3. Phase Ib: Patients who received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, and other anti-tumor treatment within 4 weeks before the first administration, except for the following: Nitrosourea or mitomycin C was received within 6 weeks before the first administration; Oral fluoropyrimidines and small molecule targeted drugs within 2 weeks or 5 half-lives of the drug (whichever is longer) prior to the first administration.Chinese proprietary medicines with anti-tumor indications were received within 2 weeks before the first administration.
* 4. Receipt of other non-marketed investigational drugs or treatments within 4 weeks before the first administration.
* 5. Patients who have received systemic glucocorticoids (prednisone > 10 mg/day or equivalent doses of similar drugs) or other immunosuppressive agents within 14 days before the first administration; exclude the following conditions: topical, ophthalmic, intra-articular, intranasal or inhaled corticosteroid therapy; short-term use of glucocorticoid for preventive treatment (for example, prevention of contrast agent allergy).
* 6.The adverse reactions of previous anti-tumor treatments have not recovered to CTCAE 5.0 grade evaluation ≤1 grade.Or the relevant provisions of the selection criteria (except for the toxicity that the researcher judges to have no safety risk).
* 7. Patients who have undergone major organ surgery (excluding needle biopsy) or have significant trauma within 4 weeks before the first administration, or require elective surgery during the trial.
* 8.Previously received allogeneic hematopoietic stem cell transplantation or organ transplantation.
* 9. Brain parenchymal metastasis or meningeal metastasis with clinical symptoms.
* 10. active infection and currently needs intravenous anti-infection treatment.
* 11. immunodeficiency disease, including HIV antibody positive.
* 12. Active hepatitis B (HBsAg positive and HBV-DNA positive or above normal) Limit), active hepatitis C (hepatitis C virus antibody positive and HCV RNA positive Or greater than the upper limit of normal value).
* 13.Vaccinated with any live vaccine within 4 weeks before the first use of the study drug.
* 14. Hypersensitivity to any antibody drugs (NCI CTCAE 5.0 grade evaluation ≥3 Grade), or active ingredients or inactive excipients of research drugs and PD-1/PD-L1 inhibitors.
* 15.With serious and uncontrollable lung diseases (severe infectious pneumonia, interstitial lung disease Etc.); Or other serious effects that may interfere with the detection or treatment of drug-related pulmonary toxicity. Moderate and severe lung diseases with respiratory function.
* 16. History of serious cardiovascular and cerebrovascular diseases, including but not limited to: Patients with severe cardiac rhythm or conduction abnormalities, such as arrhythmia requiring clinical intervention, second-degree to third-degree atrioventricular block; QT interval (QTcF) corrected by Fridericia's method > 470 ms (see Appendix 9 for calculation formula); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 and above cardiovascular and cerebrovascular events within 6 months prior to the first dose; Patients with heart failure with cardiac function class ≥ II according to New York Heart Association (NYHA) (see Appendix 4) or Left Ventricular Ejection Fraction (LVEF) < 50%; Clinically uncontrolled hypertension.
* 17. Patients who currently have active or have had autoimmune diseases that may have recurrence (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for clinically stable autoimmune thyroid diseases, type I Diabetics.
* 18. Suffering from other malignant tumors within 5 years before the start of drug administration, except for the following cases: Malignant tumor that can be expected to be cured after treatment (including but not limited to fully treated thyroid gland) cervical carcinoma in situ, basal or squamous cell skin cancer or breast treated by radical surgery. Ductal carcinoma in situ, etc.).
* 19. Clinically uncontrolled effusion in the third space, which is not suitable for enrollment based on the investigator's judgment.
* 20. Known alcohol or drug dependence.
* 21. Patients with mental disorders or poor compliance.
* 22. Women who are pregnant or breastfeeding.
* 23. The subject has a history of other serious systemic diseases or other reasons that make the subject unsuitable for this clinical study in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and SAEs (Phase Ib) | 3 months after end event visit
  To investigate the safety characteristics.
Dose limiting toxicities (DLTs) (Phase Ib) | 21 days after first dose
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D).
PFS in dose expansion (Phase II) | Baseline through up to 2 years or until disease progression
  To explore the clinical effectiveness. Tumor response based on RECIST 1.1.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Cmax (Phase Ib) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Cmax) following single dose.
Pharmacokinetic (PK) Cmin (Phase Ib) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Cmin) following single dose.
Pharmacokinetic (PK) Tmax (Phase Ib) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Tmax) following single dose.
Pharmacokinetic (PK) AUC 0-t (Phase Ib) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUC 0-t) following single dose.
Pharmacokinetic (PK) AUC 0-∞ (Phase Ib) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUC 0-∞) following single dose.
Pharmacokinetic (PK) Vd (Phase Ib) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Vd) following single dose.
Pharmacokinetic (PK) t1/2 (Phase Ib) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (t1/2) following single dose.
Pharmacokinetic (PK) λz (Phase Ib) | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (λz) following single dose.
Pharmacokinetic (PK) Css,max | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,max) following multiple dose.
Pharmacokinetic (PK) Css,min | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,min) following multiple dose.
Pharmacokinetic (PK) Css,av | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,av) following multiple dose.
Pharmacokinetic (PK) AUCss | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUCss) following multiple dose.
Pharmacokinetic (PK) CKss | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (CLss) following multiple dose.
Pharmacokinetic (PK）Vss | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Vss) following multiple dose.
Pharmacokinetic (PK) R | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (R) following multiple dose.
Pharmacokinetic (PK) DF | Day1，2，3，4，6，7，11，14，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (DF) following multiple dose.
Objective response rate (ORR) in dose escalation (Phase Ib) | Baseline through up to 2 years or until disease progression
  Tumor response based on RECIST 1.1.
Incidence of adverse events (AEs) and SAEs (Phase Ib) | 3 months after end event visit
  To investigate the safety characteristics.
Immunogenicity of IAH0968 (Phase Ib) | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IAP0971.(Phase Ib)
ORR (Phase Ⅱ) | Baseline through up to 2 years or until disease progression
  ORR as assessed using RECIST 1.1.
Overall survival (OS) (Phase II) | Baseline through up to 2 years or until disease progression
  OS as assessed using RECIST 1.1.
Disease control rate (DCR) (Phase II) | Baseline through up to 2 years or until disease progression
  DCR as assessed using RECIST 1.1.
Incidence of adverse events (AEs) and SAEs (Phase II) | 3 months after end event visit
  To investigate the safety characteristics.
Immunogenicity of IAH0968 (Phase II) | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IAP0971.(Phase II)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
we donot share.